CLINICAL TRIAL: NCT02846428
Title: An Open-Label, Multicenter, Randomized, Phase II Study to Evaluate the Efficacy and Safety of Two Combination Dose Regimens: Capecitabine + Epirubicin + Cyclophosphamide (CEX) Versus 5-FU + Epirubicin + Cyclophosphamide (FEC 100) as Neoadjuvant Therapy in Females Presenting With Operable Breast Cancer
Brief Title: To Evaluate the Efficacy and Safety of Capecitabine Prior to Surgery in Women With Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML16986
Record Dates: First submitted 2016-07-25; First posted 2016-07-27 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fluorouracil; Capecitabine; Cyclophosphamide; Docetaxel; Epirubicin

ARMS (2):
- 5-Fluorouracil + Epirubicin + Cyclophosphamide (Active Comparator): Neoadjuvant treatment (Period 1): Participants will receive 4 cycles (cycle length = 21 days) of 5-FU + epirubicin + cyclophosphamide. Surgery will be performed 5 (+/- 1) weeks after the last cycle. Adjuvant treatment (Period 2): Participants will receive 4 cycles (cycle length = 21 days) of docetaxel.
  Interventions: Drug: 5-Fluorouracil; Drug: Cyclophosphamide; Drug: Docetaxel; Drug: Epirubicin
- Capecitabine + Epirubicin + Cyclophosphamide (Experimental): Neoadjuvant treatment (Period 1): Participants will receive 4 cycles (cycle length = 21 days) of capecitabine + epirubicin + cyclophosphamide. Surgery will be performed 5 (+/- 1) weeks after the last cycle. Adjuvant treatment (Period 2): Participants will receive 4 cycles (cycle length = 21 days) of docetaxel.
  Interventions: Drug: Capecitabine; Drug: Cyclophosphamide; Drug: Docetaxel; Drug: Epirubicin

INTERVENTIONS:
Drug: 5-Fluorouracil — 5-FU will be administered at 500 mg/m^2 by short IV infusion on Day 1 of each 21-day cycle during neoadjuvant treatment period for 4 cycles.
  Arms: 5-Fluorouracil + Epirubicin + Cyclophosphamide
Drug: Capecitabine — Capecitabine will be administered at 900 mg/m^2 orally twice daily on Days 1-14 of each 21-day cycle for 4 cycles during neoadjuvant treatment period.
  Other Names: Xeloda
  Arms: Capecitabine + Epirubicin + Cyclophosphamide
Drug: Cyclophosphamide — Cyclophosphamide will be administered at 500 mg/m^2 by short IV infusion on Day 1 of each 21-day cycle for 4 cycles during neoadjuvant treatment period.
Drug: Docetaxel — Docetaxel will be administered at 100 mg/m^2 by IV infusion on Day 1 of each 21-day cycle for 4 cycles during adjuvant treatment period.
Drug: Epirubicin — Epirubicin will be administered at 100 mg/m^2 by short IV infusion on Day 1 of each 21-day cycle for 4 cycles during neoadjuvant treatment period.

SUMMARY:
This study will evaluate the efficacy and safety of treatment with oral capecitabine or intravenous (IV) 5-fluorouracil (5-FU), in combination with epirubicin and cyclophosphamide, prior to surgery in participants with breast cancer. The participants will receive 4 cycles of neoadjuvant Capecitabine + Epirubicin + Cyclophosphamide (CEX) or 5-FU + Epirubicin + Cyclophosphamide (FEC 100) chemotherapy during first treatment period (Period 1, Days 1-85). After 4-6 weeks of the fourth cycle of neoadjuvant chemotherapy (Day 120 +/- 7 days), breast surgery with regional lymph node dissection will be performed, followed within a maximum of 6 weeks by the second treatment period (Period 2, Days 1 to 85) when participants in both study arms will receive 4 cycles of adjuvant docetaxel 100 milligrams per meter square (mg/m^2) by IV infusion on Day 1 of each 21-day cycle. Upon completion of the second treatment period, participants will enter the post-treatment follow-up period which will last for 5 years from the initial date of participant randomization. During this period participants will be evaluated once a year on the anniversary date of randomization.

ELIGIBILITY:
Inclusion Criteria:

* Females with a unilateral, non-inflammatory, non-multicentric, non-metastatic breast adenocarcinoma, not considered candidates for conservative management, and whose diagnosis had been histologically confirmed as T2-3, N0-1, M0 according to the tumor-nodes-metastasis (TNM) classification
* Clinically or radiologically measurable lesion (in 2 dimensions)
* Eastern Cooperative Oncology Group (ECOG) performance Status less than equal to (<=) 1

Exclusion Criteria:

* Females presenting with brain metastases or a neurological or psychiatric disorder which could interfere with proper treatment compliance
* Previous radiotherapy, chemotherapy, or hormonal therapy for breast cancer
* Previous history of a malignancy in last 5 years other than cutaneous basal cell carcinoma or carcinoma in situ of the uterine cervix
* Serious concomitant infection
* Pregnant or lactating females

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2004-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with pathological complete tumor response Assessed by Expert Blinded Independent Review according to the Sataloff classification\n | Day 120 +/- 7 days

SECONDARY OUTCOMES:
Percentage of participants with pathological complete tumor response Assessed by Investigator according to the Sataloff classification | Day 120 +/- 7 days
Percentage of participants with breast conserving surgery | Day 120 +/- 7 days
Percentage of participants with objective clinical response, assessed by World Health Organization (WHO) criteria | Week 15
Percentage of participants with clinical response, assessed by WHO criteria | Week 15
Percentage of participants with disease progression, assessed by WHO criteria | Baseline up to 29 +/- 1 weeks
Percentage of participants with abnormalities in bilateral mammography | Day 85
Percentage of participants who died | Baseline up to 29 +/- 1 weeks
Percentage of participants with abnormal left ventricular ejection fraction (LVEF) | Days 1-85
Percentage of participants with abnormal liver ultrasound | Days 1-85
Percentage of participants with abnormal Chest X-Ray | Days 1-85
Overall survival | Baseline up to 5 years
Disease free survival, according to WHO criteria | Baseline up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (21):
- France (21):
  - Bayonne
  - Béziers
  - Bourg-en-Bresse
  - Colmar
  - Dijon
  - Hyères
  - La Tronche
  - Le Mans
  - Limoges
  - Lyon
  - Marseille
  - Montbéliard
  - Montfermeil
  - Nice
  - Nîmes
  - Paris
  - Pierre-Bénite
  - Saint-Herblain
  - Strasbourg
  - Toulouse
  - Vannes